CLINICAL TRIAL: NCT03875105
Title: The Investigation of Daily Living Activities and Exercise Capacity in Lipid Storage Diseases
Brief Title: Daily Living Activities and Exercise Capacity in Lipid Storage Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associated Proffesor, Istanbul University
Other Study IDs: 2018/24-13
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Lipid Storage Disease
Keywords: exercise capacity; activities of daily living
MeSH Terms: conditions — Lipidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lipid Storage Diseases (LSD) is a group of metabolic diseases that are manifested by exercise intolerance or muscle weakness, sometimes accompanied by systemic findings, which develop in some stages of muscle contraction due to necessary lipid transfer or destruction pathways. Exercise intolerance in LSD can limit not only physical activity but also daily activities. In the literature, no study evaluated the activities of daily living in patients with LSD. The aim of this study was to investigate the effect of exercise capacity and daily living activities on the clinical features of LSD patients.

DETAILED DESCRIPTION:
Pulmonary functions are affected negatively in Lipid Storage Diseases (LSD). It was shown that respiratory muscle strength and peak cough flow decreased in these cases. Other respiratory system problems can be listed as; diaphragmatic dysfunction, hypoxemia, and hypercapnia. Routine evaluation of respiratory function in LSD is recommended. A limited number of studies have shown that exercise tolerance is limited by the blockage of fat oxidation on the basis of muscle weakness and fatigue in LSD. Although the assessment of exercise capacity is also an important indicator of heart-lung capacity monitoring, exercise capacity is not routinely measured in patients with LSD. Exercise intolerance can limit not only physical activity but also daily activities. In the literature, the investigator's did not find any study evaluating the activities of daily living in patients with LSD. The aim of this study was to investigate the effect of exercise capacity and daily living activities on the clinical features of LSD patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Lipid storage disease clinically and histopathologically.

Exclusion Criteria:

* Severe pulmonary parenchymal disease,
* Cardiac problems
* Renal or hepatic dysfunction
* Uncontrolled hypothyroidism
* Acute infection
* Malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 25 patients who were diagnosed with Lipid Storage Disease at Istanbul University Istanbul Medical Faculty Neurology and Chest Diseases Departments will be invited to the study. The study will be continued in Istanbul University, Istanbul Faculty of Medicine, Department of Chest Diseases.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-09-02 (Estimated); Primary Completion 2024-09-04 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking test | 1 day
  Exercise capacity will be evaluated with 6 minutes walking test

SECONDARY OUTCOMES:
Activity limitation (ACTIVLIM) questionnaire | 1 day
  Activities of daily living will be evaluated Activlim questionnaire. The questionnaire is consists of 22 questions. Minimum score is 0 and total score is 88. Higher scores indicate worse conditions.
Rivermead mobility index | 1 day
  Mobility will be evaluated with Rivermead mobility index. The questionnaire consists of 14 questions. Minimum score is 0, maximum score is 15. Higher scores indicate better conditions.
Hand held dinamometer | 1 day
  Hand held dinamometer will be used for the measurement of upper and lower muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Goksen Kuran Aslan, Assoc.Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bingol Z, Tekce HD, Sagcan G, Serdaroglu P, Kiyan E. Pulmonary functions and sleep-related breathing disorders in lipid storage disease. Sleep Breath. 2018 Dec;22(4):1137-1142. doi: 10.1007/s11325-018-1647-1. Epub 2018 Mar 1. PMID 29497949